CLINICAL TRIAL: NCT05211960
Title: Effects of a Mindfulness App for Outpatients Waitlisted for Psychological Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Lena Quilty, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 088/2021
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Mental Disorder
Keywords: mindfulness; digital health
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Masking Description: All participants will be recruited knowing that a mindfulness app will be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): AmDTx is a mindfulness-based meditation app that includes lessons, interactive exercises, and additional in-app features to practice mindfulness. Participants will receive a premium account for 1 year; the current study will evaluate outcomes over 3 months. The intervention will be delivered concurrently with treatment as usual which includes standard psychosocial care as participants are referred to their respective programs.
  Interventions: Behavioral: Mindfulness-based meditation

INTERVENTIONS:
Behavioral: Mindfulness-based meditation — AmDTx is a mindfulness-based meditation app that includes lessons, interactive exercises, and additional in-app features to practice mindfulness.
  Other Names: AmDTx

SUMMARY:
The purpose of this study is to evaluate a mindfulness-based meditation app provided to outpatients (or community participants) who are waitlisted for standard psychological care for mental health or substance use concerns.

DETAILED DESCRIPTION:
This project aims to provide a previously validated mindfulness meditation app to up to 200 adults waitlisted for psychological services in a psychiatric hospital setting or in the broader community. Outpatients (or community participants) who have been referred to and waitlisted for treatment for their mood, anxiety, alcohol, and/or substance use concerns, will be offered access to the digital intervention for 1 year. We will follow participants for 3 months to evaluate usability and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Fluency in English
3. Understanding and willingness to comply with study requirements
4. Waitlisted for outpatient psychosocial programming at CAMH (or psychosocial programming in the community)
5. Smartphone or tablet capable of downloading and running the mindfulness app.

Exclusion Criteria:

1. Any known practical factor that would preclude participation (e.g., extended absences)
2. Acute psychiatric (e.g., acute suicidality, psychosis) or serious medical condition that precludes participation in this study.
3. Participation in another treatment/intervention study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS 2.0) Short Form | 30 days
  Level of functional disability in the past month across six subdomains. Minimum score: 0, Maximum score: 48. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) Depression Subscale | 14 days
  Level of depressive symptoms over the past two weeks. Minimum score: 0, Maximum score: 27. Higher scores mean worse outcome.
Generalized Anxiety Disorder 7 (GAD-7) Scale | 14 days
  Level of generalized anxiety symptoms over the past two weeks. Minimum score: 0, Maximum score: 21. Higher scores mean worse outcome.
Five Factor Mindfulness Questionnaire, Short Form (FFMQ-SF) | 30 days
  Measure of five core mindfulness skills over the past month (15 items). Minimum score: 15, Maximum score: 75. Higher scores mean greater dispositional mindfulness (good outcome).
Philadelphia Mindfulness Scale | 30 days
  Measure of mindful acceptance and awareness over the past month (20 items). Minimum score: 20, Maximum score: 100. Higher scores mean greater dispositional mindfulness (good outcome).
Perceived Stress Scale | 30 days
  Well-validated measure of perceived stress over the past month (10 items). Minimum score: 0, Maximum score: 40. Higher scores mean greater perceived stress (worse outcome).
Ruminative Response Scale, Short Form (Treynor & Nolen-Hoeksema, 2003) | 30 days
  Measure of ruminative thought patterns over the past 30 days using 10 items. Minimum score: 10, Maximum score: 40. Higher scores mean greater tendency to ruminate (worse outcome).
Repetitive Thinking Questionnaire | 30 days
  Measure of negative repetitive thought patterns over the past 30 days using 10 items. Minimum score: 10, Maximum score: 50. Higher scores mean greater tendency to experience repetitive thinking (worse outcome).
Penn State Worry Questionnaire | 30 days
  Measure of worry and rumination over the past 30 days using 16 items. Minimum score: 16, Maximum score: 80. Higher scores mean greater tendency to worry (worse outcome).
Work Productivity and Activity Impairment | 30 days
  Measure of disruption to work and activities because of mental health symptoms in the past month using 5 items. Scores vary as the scale utilizes open response options to some questions. Higher scores generally indicate more impairment to productivity.
Treatment Acceptability Questionnaire (Hunsley, 1992) | 30 days
  Assesses the patient's perception of the treatment as useful, helpful, and effective using 6 items. Minimum score: 6, Maximum score: 42. Higher scores indicate greater acceptability.
MHealth App Usability Questionnaire | 30 days
  An 18-item measure of the ease of use, acceptability as a treatment, and satisfaction. Minimum score: 18, Maximum score: 126. Higher scores indicate greater usability and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lena C. Quilty, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Campbell Family Mental Health Research Institute, CAMH, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca